CLINICAL TRIAL: NCT00293033
Title: A Double-blind, Placebo Controlled Evaluation of the Efficacy, Safety and Tolerability of BEMA™ Fentanyl in the Treatment of Breakthrough Pain in Cancer Subjects
Brief Title: Study of BEMA™ Fentanyl in the Treatment of Breakthrough Pain in Cancer Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FEN-201
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Pain; Cancer
Keywords: Breakthrough Pain in Patients with Cancer
MeSH Terms: conditions — Pain; Neoplasms | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: BEMA™; Drug: Placebo
- BEMA™ Fentanyl (Experimental): BioErodible MucoAdhesive (BEMA) Fentanyl
  Interventions: Drug: BEMA™

INTERVENTIONS:
Drug: BEMA™ — BioDelivery Sciences International, Inc. (BDSI) has developed BioErodible MucoAdhesive (BEMA) Fentanyl, an alternative product to OTFC that does not require the subject to continuously paint the inside of the mouth with the dosage form. The BDSI product is a small soluble film that is placed against the mucosal membrane inside the mouth. The mucoadhesive polymers in the film readily adhere to the mucosal membrane (within 5 seconds) when moistened. The components of the film are water soluble, so the entire dosage form dissolves within 30 minutes of application.
  Other Names: Onsolis (fentanyl buccal soluble film)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of BEMA Fentanyl (Onsolis) at any dose in the management of breakthrough pain in cancer subjects on background opioid therapy. The standard of care for these breakthrough pain episodes is a rapid onset, short acting analgesic with minimal associated sleepiness. Oral morphine, oxycodone and hydromorphone are routinely used, but because of slow and variable oral absorption, the pain control is not the best with these products. Oral transmucosal fentanyl citrate (OTFC) has been used successfully in treating breakthrough pain episodes associated with cancer. OTFC is a lozenge of fentanyl on a stick and is administered by continuously swabbing the interior of the subject's mouth until the product is dissolved (approximately 15 to 30 minutes). The buccal route of administration avoids the delay and variability associated with oral absorption.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, multiple cross-over study. Eligible subjects will be treated with open label BEMA fentanyl over a period of up to two weeks. Doses will be titrated upward, starting at 200 μg, until a dose is identified that produces satisfactory pain relief for at least 2 episodes. Those subjects who identify a dose of BEMA fentanyl that produces satisfactory relief of breakthrough pain episodes will enter the double-blind, placebo controlled period of the trial. They will receive 3 placebo doses and 6 BEMA fentanyl doses in a random sequence per randomization schedule.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-lactating female. A female of child-bearing potential is eligible to participate in this study if she is using an acceptable method of birth control.
* 18 years or older
* Patient must have pain associated with cancer or cancer treatment.
* Patient must be on a stable current regimen of oral opioids equivalent to 60 - 1000 mg/day of oral morphine or 50 - 300 µg/hr of transdermal fentanyl (e.g. oxycodone 30 mg, methadone 20 mg, and hydromorphone 7.5 mg).
* Regularly experiences 1 - 4 breakthrough pain episodes per day that require additional opioids for pain control
* At least partial relief of breakthrough pain by use of opioid therapy
* Subject must be able to self-administer the study medication correctly.
* Subject must be willing and able to complete the electronic diary card with each pain episode.
* Signed consent must be obtained at screening prior to any procedures being performed.

Exclusion Criteria:

* Psychiatric/cognitive or neurological impairment that would limit the subject's ability to understand or complete the diary
* Cardiopulmonary disease that, in the opinion of the investigator, would significantly increase the risk of respiratory depression
* Recent history or current evidence of alcohol or other drug substance (licit or illicit) abuse
* Rapidly escalating pain that the investigator believes may require an increase in the dosage of background pain medication during the study
* Moderate (Grade 3) to severe (Grade 4) mucositis (Subjects with less than moderate mucositis are permitted and must be instructed to not apply the BEMA disc at a site of inflammation.)
* Strontium 89 therapy within the previous 6 months
* Any other therapy prior to the study that the investigator considers could alter pain or the response to pain medication.
* Use of an investigational drug within 4 weeks preceding this study
* History of hypersensitivity or intolerance to fentanyl
* Regularly more than 4 episodes per day
* Eastern Cooperative Oncology Group (ECOG) performance status of 4 or 5
* Subject is pregnant, actively trying to become pregnant, breast feeding or not using adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Finn, PharmD, Study Chair — BioDelivery Sciences International
Locations (1):
- PPD Development, Wilmington, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24FEB2006 to 14MAR2007
Pre-assignment Details: During the open-label titration period, subjects were treated with Onsolis at escalating doses (200, 400, 600, 800, and 1200 μg) over a period of up to two weeks until subjects identified a dose that produced satisfactory pain relief for at least two episodes.
Groups:
- Onsolis: Subjects were administered BEMA™ Fentanyl at escalating doses (200, 400, 600, 800, and 1200 μg) in Titration period. During the double-blind period, subjects were randomly assigned to a sequence of active and placebo discs. Each subject acted as his or her own control. For each subject, the sequencing of the placebo and BEMA™ Fentanyl discs was random.
Period: Open-label Titration Period
Arm/Group | Onsolis
Started | 151 (152 subjects enrolled; 151 subjects received at least one dose of study drug)
Completed | 82
Not Completed | 69
Not completed — Adverse Event | 10
Not completed — Death | 3
Not completed — Lack of Efficacy | 5
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 22
Not completed — Noncompliance and other | 27
Period: Double-blind Treatment Period
Arm/Group | Onsolis
Started | 82 (82 randomized; 1 didn't take double-blind drug; 1 didn't report a pain assessment within 30 minutes)
Completed | 70
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 4
Not completed — Noncompliance | 4

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Onsolis: Includes all subjects and all dose levels
Arm/Group | Onsolis
Number analyzed (Participants) | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 104
  >=65 years | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 131
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 151
Female reproductive status [Count of Participants; unit: Participants]
  Post-menopausal | 43
  Sterile | 38
  Potentially able to bear children | 3
  Male | 67
Height (inches) [Mean (Standard Deviation); unit: Inches] | 66.4 (3.86)
Weight (pounds) [Mean (Standard Deviation); unit: pounds] | 160.89 (42.011)

OUTCOME MEASURES:

1. Primary Outcome: Summary of Pain Intensity Differences (SPID)
Description: Pain intensity (using an 11-point [0 = no pain to 10 = worst pain] numeric scale) was recorded at 0, 5, 10, 15, 30, 45, and 60 minutes after dosing. Pain intensity difference (PID) was defined as the baseline pain score minus the pain score of each time point. The primary endpoint was the Summary of Pain Intensity Differences at 30 minutes after dosing (SPID 30) in ITT population for Onsolis versus placebo during double-blind period of study. SPID was calculated as a weighted sum of the PID of all time points at or before time point of interest.Range of possible SPID values is
  -10X time point (minutes) to 10X time point (minutes). Higher value indicates a better outcome.
Time Frame: 0-30 minutes
Population: In double-blind period, subjects received 3 doses placebo and 6 doses Onsolis. Mean SPID of Onsolis episodes and mean SPID of placebo episodes are calculated per subject and are used in analysis.Missing data were imputed on an episode-by-episode basis by carrying forward last observed data value (last observation carried forward [LOCF]).
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Units Other Than Participants: Breakthrough Pain (BTP) Episodes
Groups:
- Onsolis: BioErodible MucoAdhesive (BEMA) Fentanyl
- Placebo: Placebo Disc
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (Breakthrough Pain (BTP) Episodes) | 394 | 197
Score on a scale | 47.9 (3.87) | 38.1 (4.3)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; The SPID was analyzed using a mixed model of repeated measures with fixed effects for treatment, pooled site, and a random effect for subjects; Mean Difference (Final Values) = 9.74, 95% CI 2-sided [3.31 to 16.18], Standard Error of Mean 3.28 — Onsolis minus placebo

2. Secondary Outcome: SPID
Description: Pain intensity (using an 11-point [0 = no pain to 10 = worst pain] numeric scale) was recorded at 0, 5, 10, 15, 30, 45, and 60 minutes after dosing. Pain intensity difference (PID) was defined as the baseline pain score minus the pain score of each time point. The primary endpoint was the Summary of Pain Intensity Differences at 30 minutes after dosing (SPID 30) in ITT population for Onsolis versus placebo during double-blind period of study. SPID was calculated as a weighted sum of the PID of all time points at or before time point of interest.Range of possible SPID values is -10X time point (minutes) to 10X time point (minutes). Higher value indicates a better outcome.SPID was calculated as a weighted sum of the pain intensity difference of all time points at or before the time point of interest.
Time Frame: 0-5 minutes
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 361 | 176
Scores on a scale | 1.8 (0.30) | 1.5 (0.36)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.440, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.40 to 0.91], Standard Error of Mean 0.33

3. Secondary Outcome: SPID
Description: as for outcome 2
Time Frame: 0-10 minutes
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 379 | 184
Scores on a scale | 5.9 (0.80) | 4.9 (0.90)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.179, Mixed Models Analysis; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [-0.44 to 2.33], Standard Error of Mean 0.70

4. Secondary Outcome: SPID
Description: as for outcome 2
Time Frame: 0-15 minutes
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 382 | 194
Scores on a scale | 12.8 (1.47) | 10.4 (1.61)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.047, Mixed Models Analysis; Mean Difference (Final Values) = 2.32, 95% CI 2-sided [0.04 to 4.61], Standard Error of Mean 1.16

5. Secondary Outcome: SPID
Description: as for outcome 2
Time Frame: 0-45 minutes
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 382 | 194
Scores on a scale | 90.5 (6.63) | 70.8 (7.41)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 19.68, 95% CI 2-sided [8.50 to 30.86], Standard Error of Mean 5.70

6. Secondary Outcome: SPID
Description: as for outcome 2
Time Frame: 0-60 minutes
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 382 | 194
Scores on a scale | 138.0 (9.41) | 106.0 (10.58)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 31.98, 95% CI 2-sided [15.85 to 48.12], Standard Error of Mean 8.23

7. Secondary Outcome: PID
Description: Pain intensity (using an 11-point [0 = no pain to 10 = worst pain] numeric scale) was recorded at 0, 5, 10, 15, 30, 45, and 60 minutes after dosing. Pain intensity difference (PID) was defined as the baseline pain score minus the pain score of each time point.
Time Frame: 5 minutes after dosing
Population: During the double-blind period, subjects received 3 doses of placebo and 6 doses of Onsolis.
  All efficacy analyses were conducted using the intent-to-treat (ITT) population.
  Last observation carried forward (LOCF) is used to impute missing data or data after rescue medication usage.
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 361 | 176
Scores on a scale | 0.3 (0.04) | 0.3 (0.06)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.517, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: PID
Description: as for outcome 7
Time Frame: 10 minutes after dosing
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 379 | 184
Scores on a scale | 0.8 (0.07) | 0.7 (0.08)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.458, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: PID
Description: as for outcome 7
Time Frame: 15 minutes after dosing
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 382 | 194
Scores on a scale | 1.4 (0.09) | 1.2 (0.10)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.223, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: PID
Description: as for outcome 7
Time Frame: 30 minutes after dosing
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 394 | 197
Scores on a scale | 2.5 (0.11) | 1.9 (0.14)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.015, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: PID
Description: as for outcome 7
Time Frame: 45 minutes after dosing
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 404 | 198
Scores on a scale | 3.0 (0.13) | 2.3 (0.17)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: PID
Description: as for outcome 7
Time Frame: 60 minutes after dosing
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 408 | 198
Scores on a scale | 3.3 (0.13) | 2.4 (0.18)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Pain Relief
Description: Pain relief (PR) is measured using a 5-point categorical scale (0=no relief to 4=complete relief) at 5, 10, 15, 30, 45, and 60 minutes after taking the study medication or until rescue.
Time Frame: 5 minutes after dosing
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 361 | 176
Scores on a scale | 0.4 (0.04) | 0.4 (0.06)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.193, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Pain Relief
Description: as for outcome 13
Time Frame: 10 minutes after dosing
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 379 | 184
Scores on a scale | 0.8 (0.05) | 0.7 (0.06)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.113, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Pain Relief
Description: as for outcome 13
Time Frame: 15 minutes after dosing
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 382 | 194
Scores on a scale | 1.1 (0.05) | 1.0 (0.07)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.192, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Pain Relief
Description: as for outcome 13
Time Frame: 30 minutes after dosing
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 394 | 197
Scores on a scale | 1.7 (0.05) | 1.3 (0.08)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Pain Relief
Description: as for outcome 13
Time Frame: 45 minutes after dosing
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 404 | 198
Scores on a scale | 1.9 (0.06) | 1.5 (0.09)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Pain Relief
Description: as for outcome 13
Time Frame: 60 minutes after dosing
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 409 | 198
Scores on a scale | 2.1 (0.06) | 1.6 (0.09)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Total Pain Relief
Description: Total Pain Relief (TOTPAR) is calculated as the weighted sum of the pain relief (PR) of all time points at or prior to the time point of interest.Pain relief (PR) is measured using a 5-point categorical scale (0=no relief to 4=complete relief)compared to baseline (pre-dose)
Time Frame: 5 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 361 | 176
Scores on a scale | 2.2 (0.21) | 1.8 (0.28)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.157, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Total Pain Relief
Description: Total Pain Relief (TOTPAR) is calculated as the weighted sum of the pain relief (PR) of all time points at or prior to the time point of interest. Pain relief (PR) is measured using a 5-point categorical scale (0=no relief to 4=complete relief)compared to baseline (pre-dose)
Time Frame: 10 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 379 | 184
Scores on a scale | 6.1 (0.40) | 5.2 (0.54)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.278, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Total Pain Relief
Description: as for outcome 20
Time Frame: 15 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 382 | 194
Scores on a scale | 11.6 (0.62) | 9.8 (0.82)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.062, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Total Pain Relief
Description: as for outcome 20
Time Frame: 30 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 394 | 197
Scores on a scale | 36.1 (1.30) | 29.5 (1.79)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Total Pain Relief
Description: as for outcome 20
Time Frame: 45 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 404 | 198
Scores on a scale | 64.2 (2.05) | 52.3 (2.93)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Total Pain Relief
Description: as for outcome 20
Time Frame: 60 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: BTP Episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (BTP Episodes) | 409 | 198
Scores on a scale | 94.8 (2.84) | 76.0 (4.16)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Subject Overall Satisfaction With Study Drug
Description: Subjects evaluated their overall satisfaction with study drug at the time rescue medication was consumed or at the 60-minute time point using a 5-point categorical scale (0 = poor, 1 = fair, 2 = good, 3 = very good, and 4 = excellent).
Time Frame: 60 minutes or at time of rescue medication use
Population: All efficacy analyses were conducted using the intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: Subject Overall Satisfaction
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
Number analyzed (Subject Overall Satisfaction) | 359 | 174
Scores on a scale | 2.0 (0.06) | 1.5 (0.10)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Percentage of Pain Free Episodes
Description: A pain free episode is one with 0 pain intensity at the specified time point. Percentage of episodes that are pain-free per subject is analyzed.
Time Frame: 5 minutes
Population: During the double-blind period, subjects received 3 doses of placebo and 6 doses of Onsolis.
  All efficacy analyses were conducted using the intent-to-treat (ITT) population, however, only available data is summarized here.
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 74
percentage of episodes | 1.0 (0.73) | 1.4 (1.37)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 1.000, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Percentage of Pain Free Episodes
Description: as for outcome 26
Time Frame: 10 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percentage of episodes
Groups:
- Onsolis: BioErodible MucoAdhesive (BEMA) Fentanyl - Includes all subjects and all dose levels.
- Placebo: Placebo Disc - Includes all subjects and all dose levels.
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 74
percentage of episodes | 1.0 (0.72) | 1.4 (1.35)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 1.000, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Percentage of Pain Free Episodes
Description: as for outcome 26
Time Frame: 15 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 74
percentage of episodes | 2.3 (1.02) | 2.0 (1.48)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.563, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Percentage of Pain Free Episodes
Description: as for outcome 26
Time Frame: 30 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 76
percentage of episodes | 5.3 (1.57) | 4.4 (1.88)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.498, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Percentage of Pain Free Episodes
Description: as for outcome 26
Time Frame: 45 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 76
percentage of episodes | 10.5 (2.34) | 6.4 (2.27)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.077, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Percentage of Pain Free Episodes
Description: as for outcome 26
Time Frame: 60 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 78 | 76
percentage of episodes | 14.2 (2.62) | 9.6 (2.90)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.031, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: Episodes With at Least 50% Decreases in Pain
Description: Number of episodes where the total pain score has at least a 50% reduction from baseline.
Time Frame: 15 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 75
episodes | 14.9 (2.81) | 14.7 (3.35)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.963, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: Episodes With at Least 50% Decreases in Pain
Description: Number of episodes where the total pain score has at least a 50% reduction from baseline.
Time Frame: 30 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 76
episodes | 32.8 (3.78) | 24.1 (3.87)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: Episodes With at Least 50% Decreases in Pain
Description: Number of episodes where the total pain score has at least a 50% reduction from baseline.
Time Frame: 45 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 76
episodes | 41.1 (4.11) | 30.5 (4.10)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Episodes With at Least 50% Decreases in Pain
Description: Number of episodes where the total pain score has at least a 50% reduction from baseline.
Time Frame: 60 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 78 | 76
episodes | 46.1 (4.17) | 34.0 (4.30)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Episodes With at Least 33% Decreases in Pain
Description: Number of episodes where the total pain score has at least a 33% reduction from baseline.
Time Frame: 15 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 75
episodes | 26.4 (3.55) | 21.3 (3.66)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.100, Wilcoxon (Mann-Whitney)

37. Secondary Outcome: Episodes With at Least 33% Decreases in Pain
Description: Number of episodes where the total pain score has at least a 33% reduction from baseline.
Time Frame: 30 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 76
episodes | 47.3 (4.05) | 38.2 (4.45)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.009, Wilcoxon (Mann-Whitney)

38. Secondary Outcome: Episodes With at Least 33% Decreases in Pain
Description: Number of episodes where the total pain score has at least a 33% reduction from baseline.
Time Frame: 45 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 76
episodes | 57.5 (3.93) | 46.5 (4.50)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

39. Secondary Outcome: Episodes With at Least 33% Decreases in Pain
Description: Number of episodes where the total pain score has at least a 50% reduction from baseline.
Time Frame: 60 minutes
Population: as for outcome 7
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 78 | 76
episodes | 64.3 (3.72) | 48.2 (4.51)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

40. Secondary Outcome: Episodes With Complete Pain Relief
Description: Pain relief (PR) is measured using a 5-point categorical scale (0=no relief to 4=complete relief). Percentage of episodes with complete relief per subject is analyzed where a complete pain relief episode is defined as pain relief of value 4 at the specified time point.
Time Frame: 5 minutes
Population: All efficacy analyses were conducted using the intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 76 | 73
percentage of episodes | 0.7 (0.66) | 0.7 (0.68)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 1.000, Wilcoxon (Mann-Whitney)

41. Secondary Outcome: Episodes With Complete Pain Relief
Description: Pain relief (PR) is measured using a 5-point categorical scale (0=no relief to 4=complete relief).Percentage of episodes with complete relief per subject is analyzed where a complete pain relief episode is defined as pain relief of value 4 at the specified time point.
Time Frame: 10 minutes
Population: All efficacy analyses were conducted using the intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 74
percentage of episodes | 1.0 (0.72) | 0.7 (0.68)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 1.000, Wilcoxon (Mann-Whitney)

42. Secondary Outcome: Episodes With Complete Pain Relief
Description: as for outcome 41
Time Frame: 15 minutes
Population: All efficacy analyses were conducted using the intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 75
percentage of episodes | 1.7 (0.83) | 1.3 (0.94)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.750, Wilcoxon (Mann-Whitney)

43. Secondary Outcome: Episodes With Complete Pain Relief
Description: as for outcome 40
Time Frame: 30 minutes
Population: All efficacy analyses were conducted using the intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 76
percentage of episodes | 5.4 (1.63) | 2.6 (1.33)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.032, Wilcoxon (Mann-Whitney)

44. Secondary Outcome: Episodes With Complete Pain Relief
Description: as for outcome 40
Time Frame: 45 minutes
Population: All efficacy analyses were conducted using the intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 77 | 76
percentage of episodes | 9.4 (2.18) | 6.4 (2.27)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.131, Wilcoxon (Mann-Whitney)

45. Secondary Outcome: Episodes With Complete Pain Relief
Description: as for outcome 40
Time Frame: 60 minutes
Population: All efficacy analyses were conducted using the intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 78 | 76
percentage of episodes | 12.8 (2.49) | 7.2 (2.40)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney)

46. Secondary Outcome: Rescue Medication Usage
Description: Rescue medication is medication taken if adequate pain relief is not realized within 30 minutes following application of the study drug. Percentage of episodes when rescue medication was used per subject is analyzed.
Time Frame: 28 Days
Population: All efficacy analyses were conducted using the intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: percentage of episodes
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 79 | 77
percentage of episodes | 30.0 (3.53) | 44.6 (4.38)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

47. Other Pre Specified Outcome: SPID in Neuropathic Pain Subpopulation
Description: Pain intensity (using an 11-point [0 = no pain to 10 = worst pain] numeric scale) was recorded at 0, 5, 10, 15, 30, 45, and 60 minutes after dosing. Pain intensity difference (PID) was defined as the baseline pain score minus the pain score of each time point. The primary endpoint was the Summary of Pain Intensity Differences at 30 minutes after dosing (SPID 30) in ITT population for Onsolis versus placebo during double-blind period of study. SPID was calculated as a weighted sum of the PID of all time points at or before time point of interest.Range of possible SPID values is -10X time point (minutes) to 10X time point (minutes). Higher value indicates a better outcome. SPID was calculated as a weighted sum of the pain intensity difference of all time points at or before the time point of interest for the Neuropathic pain subpopulation for relevant time points (15, 30, 45, 60 minutes). Neuropathic pain subpopulation is a subset of ITT population who have neuropathic pain at baseline.
Time Frame: 15 minutes
Population: During the double-blind period, subjects received 3 doses of placebo and 6 doses of Onsolis.
  All efficacy analyses were conducted using the intent-to-treat (ITT) population.
  Missing data were imputed on an episode-by-episode basis by carrying forward the last observed data value (last observation carried forward [LOCF]).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 23 | 22
Scores on a scale | 13.8 (2.93) | 7.8 (3.20)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; Mean Difference (Final Values) = 5.96, 95% CI 2-sided [0.92 to 11.01], Standard Error of Mean 2.57

48. Other Pre Specified Outcome: SPID in Neuropathic Pain Subpopulation
Description: as for outcome 47
Time Frame: 30 minutes
Population: as for outcome 47
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 23 | 22
Scores on a scale | 51.6 (8.05) | 31.8 (8.86)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; Mean Difference (Final Values) = 19.84, 95% CI 2-sided [5.63 to 34.04], Standard Error of Mean 7.25

49. Other Pre Specified Outcome: SPID in Neuropathic Pain Subpopulation
Description: as for outcome 47
Time Frame: 45 minutes
Population: as for outcome 47
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 23 | 22
Scores on a scale | 93.0 (14.09) | 59.7 (15.63)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; Mean Difference (Final Values) = 33.26, 95% CI 2-sided [8.32 to 58.20], Standard Error of Mean 12.72

50. Other Pre Specified Outcome: SPID in Neuropathic Pain Subpopulation
Description: as for outcome 47
Time Frame: 60 minutes
Population: as for outcome 47
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Onsolis | Placebo
Number analyzed (Participants) | 23 | 22
Scores on a scale | 137.8 (20.19) | 90.9 (22.53)
Statistical Analysis 1: Comparison: Onsolis vs Placebo; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis; Mean Difference (Final Values) = 46.88, 95% CI 2-sided [10.69 to 83.08], Standard Error of Mean 18.46

ADVERSE EVENTS:
Time Frame: A prior-treatment adverse event (AE) was defined as an AE that began before the first dose of the study drug. A treatment-emergent AE was defined as an AE that began on or after the initial dose of study medication up until the Follow-up Visit on Day 29.
Description: At each visit, after the subject had an opportunity to spontaneously mention any problems, the investigator inquired about AEs by asking the following:
  1. Have you had any (other) medical problems since your last visit/assessment?
  2. Have you taken any new medications, other than those given to you in this study, since your last visit/assessment?
Groups:
- Onsolis: All AEs were assigned to BEMA™ Fentanyl (Onsolis). Because of the multiple crossover design and the number of breakthrough pain episodes that usually occur during the day, it was likely that a subject would receive both active and placebo doses within a few hours of each other. Given the proximity of these different treatments, attempts to ascribe individual AEs to one treatment or another would be difficult, therefore, the chosen convention was to consider all AEs as occurring on active medication.
Arm/Group | Onsolis
Serious Adverse Events (participants affected / at risk) | 23/151
Other Adverse Events (participants affected / at risk) | 44/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onsolis (N=151)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Sepsis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Vaginal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onsolis (N=151)
Nausea (Gastrointestinal disorders) | 21 (21)
Vomiting (Gastrointestinal disorders) | 19 (19)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Somnolence (Nervous system disorders) | 10 (11)
Dizziness (Nervous system disorders) | 7 (7)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The oral or written use of study results by the investigator are not permitted without the express written consent from BDSI. All data resulting from this study remain property of BDSI.